CLINICAL TRIAL: NCT06663631
Title: The Safety and effiCacy of HIbernation-Like Therapy Combining recanaLization in Ischemic Stroke: a Phase 1, Dose-escalation Study
Brief Title: Study on Hibernation-like Therapy Based on Mechanical Thrombectomy
Acronym: CHILL-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, chief physician, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHILL-1
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Hibernation-like status; Reperfusion; Neuroprotection; phenothiazine; dose-escalation
MeSH Terms: conditions — Ischemic Stroke | interventions — Chlorpromazine; Promethazine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- chlorpromazine and promethazine of Very low dosage (Experimental): patients will receive C+P（chlorpromazine and promethazine ,10 mg each)at the beginning of endovascular thrombectomy.
  Interventions: Drug: chlorpromazine and promethazine; Procedure: endovascular thrombectomy; Drug: rt-PA
- chlorpromazine and promethazine of low-dosage (Experimental): patients will receive C+P（chlorpromazine and promethazine ,20 mg each)at the beginning of endovascular thrombectomy.
  Interventions: Drug: chlorpromazine and promethazine; Procedure: endovascular thrombectomy; Drug: rt-PA
- chlorpromazine and promethazine of moderate dosage (Experimental): patients will receive C+P（chlorpromazine and promethazine ,50 mg each)at the beginning of endovascular thrombectomy.
  Interventions: Drug: chlorpromazine and promethazine; Procedure: endovascular thrombectomy; Drug: rt-PA
- chlorpromazine and promethazine of high dosage (Experimental): patients will receive C+P（chlorpromazine and promethazine ,100 mg each)at the beginning of endovascular thrombectomy.
  Interventions: Drug: chlorpromazine and promethazine; Procedure: endovascular thrombectomy; Drug: rt-PA
- Placebo group (Placebo Comparator): 50 ml saline solution was delivered intravenously at the beginning of endovascular thrombectomyat a velocity of 4ml/h. The whole period of drug delivery lasts for approximately 12h.
  Interventions: Drug: Placebo group; Procedure: endovascular thrombectomy; Drug: rt-PA

INTERVENTIONS:
Drug: chlorpromazine and promethazine — C+P were diluted to 50 ml saline solution and delivered intravenously at the beginning of endovascular thrombectomyat a velocity of 4ml/h. The whole period of drug delivery lasts for approximately 12h.
  Other Names: C+P; lytic cocktail
  Arms: chlorpromazine and promethazine of Very low dosage; chlorpromazine and promethazine of high dosage; chlorpromazine and promethazine of low-dosage; chlorpromazine and promethazine of moderate dosage
Drug: Placebo group — 50 ml saline solution was set as placebo and delivered intravenously at the beginning of endovascular thrombectomyat a velocity of 4ml/h. The whole period of drug delivery lasts for approximately 12h.
  Other Names: Control group
  Arms: Placebo group
Procedure: endovascular thrombectomy — All patients that are eligible for endovascular thrombectomy will receive this surgery in aim to remove thrombus and restore reperfusion.
Drug: rt-PA — All patients that are eligible for Intravenous thrombolysis will receive 0.9mg/kg rt-PA in aim to remove thrombus and restore reperfusion
  Other Names: Intravenous thrombolysis

SUMMARY:
The goal of this clinical trial is to learn whether chlorpromazine and promethazine（C+P）is safe in Acute Ischemic Stroke（AIS) patients and determine the maximum dosage. It will also evaluate the preliminary efficacy of C+P in AIS. The main questions it aims to answer are:

What is the optimal dosage of C+P that is safe without causing adverse effects in AIS patients? What is the optimal dosage of C+P that potentially works to treat AIS? Researchers will compare C+P with placebo (saline solution without C+P) to see if C+P is safe and effective in treating Acute Ischemic Stroke.

Participants will:

Receive C+P or placebo at the same time as endovascular thrombectomy begins. Patients will be observed for 72 hours to see if there were any adverse effects related to C+P. Infarct volumes will be evaluated using Computed Tomography. Functional outcomes will be assessed at 90 days.

DETAILED DESCRIPTION:
Chlorpromazine and promethazine (C+P), due to their effort to induce a hibernation-like status, has been proved to be neuroprotective for ischemic stroke in pre-clinical experiments. However, whether it is safe and potentially effective in acute ischemic stroke (AIS) patients is currently unknown. The reason might be that the optimal dosage is not defined in AIS treatment. High dosage of C+P might result in hypotension and extrapyramidal symptoms that diminishes its neuroprotective effect. So it is essential to determine a safe and potentially dosage. Another reason might be that patients from previous clinical trials assessing the effectiveness of C+P did not receive reperfusion therapy. In this study，we plan to conduct a 6+2 dose-escalation clinical trial to determine the safety of C+P in AIS patients receiving endovascular thrombectomy. Four dosage groups of C+P will be set(10mg/20mg/50mg/100mg).A minimum of 32 patients will be involved if no drug related severe adverse event(SAE) was observed. A maximum of 64 patients will be required if one SAE is observed in each group. The current study aim to provide a basis for phase Ⅱ clinical trial to further explore the efficacy of C+P in AIS treatmment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion Criteria:

  1. Age between 18-80 years(including the critical value)
  2. Ischemic stroke with a National Institutes of Health Stroke Scale (NIHSS) score ranging from 6-20
  3. Time from last known to be well to randomization within 24h
  4. Pre-stroke Modified Rankin Scale scoring 0-1.
  5. With indications of reperfusion therapy (including intravenous thrombolysis and endovascular thrombectomy).
  6. Informed consent signed by patients or their legal relatives.
  7. CT angiography (CTA) confirmed large vessel occlusion of anterior circulation
  8. Alberta Stroke Program Early Computed Tomography Score (ASPECT) score of 6-10.
  9. initial infarct volume on CT perfusion (CTP) lesser than 70ml; a ratio of hypoperfused volume to infarcted volume greater than 1.8; absolute mismatch volume greater than 15 ml according to DEFUSE-3 trial.

Exclusion Criteria:

* Clinical Exclusion Criteria:

  1. Clinical findings suggest intracranial parenchymal hemorrhage or subarachnoid hemorrhage.
  2. Accompanied by epilepsy.
  3. Accompanied by coma or mental disorders, may interfere with neurological function assessment.
  4. History of premorbid phenothiazine allergy or contraindication.
  5. History of allergy to iodine contrast medium or anaphylactic shock
  6. Baseline blood glucose <50mg/dL (2.78mmol) or >400mg/dL (22.20mmol)

     * Acceptable fingertip blood glucose results
  7. Baseline platelet <50×109 /L
  8. Recent (i.e. within 30 days prior to randomization) history of gastrointestinal or other clinically significant bleeding; Active bleeding, abnormal clotting factors, or bleeding tendency (INR≥3 or PT≥3×ULN on anticoagulants; If the investigator believes that the subject does not have coagulation dysfunction, it is not necessary to wait for the results of the coagulation test before deciding whether to enroll.)
  9. The stroke is accompanied by fever, or there is an active infection requiring systemic treatment (such as active tuberculosis, etc.)
  10. Expected survival less than 90 days (According to the Chinese Guidelines for Early Endovascular Interventional Diagnosis and Treatment of Acute Ischemic Stroke 2022, expected survival less than 90 days is a contraindication for endovascular therapy)
  11. A history of severe cardiovascular disease, including but not limited to: uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg after standard treatment), hypotension (systolic blood pressure ≤100 mmHg after standard treatment), or pulmonary hypertension; Had unstable angina pectoris, myocardial infarction, or bypass or stent surgery within 6 months before randomization; New York Heart Association (NYHA) grade 3-4 history of chronic heart failure; Clinically significant valvular disease; Severe arrhythmias requiring treatment (except atrial fibrillation and paroxysmal supraventricular tachycardia), including QT interval ≥450ms for men and ≥470ms for women
  12. accompanied by chronic obstructive pulmonary disease（COPD）, tuberculosis, pneumonia, pneumothorax, atelectasis, pulmonary fibrosis, bronchopulmonary dysplasia, pleural effusion, acute respiratory distress syndrome, respiratory irregularity and other lung diseases
  13. Severe hepatic and renal insufficiency, including but not limited to: cirrhosis, hepatic encephalopathy, ascites, renal failure or uremia (Ccr<25ml/min), hepatorenal syndrome, etc
  14. Pregnancy or lactating women
  15. Participation in other clinical trials and have used an investigational drug or medical device
  16. Patients that may not be able to complete the study for other reasons or who the investigator believes should not be included
* Image exclusion criteria:

  1. computed tomographic angiography（CTA）/magnetic resonance angiography（MRA）/digital substraction angiography（DSA） shows excessive vascular curvature, which may hinder delivery of interventional devices
  2. Cerebrovascular inflammation is suspected based on medical history and CTA/MRA/DSA
  3. Aortic dissection is suspected based on medical history and CTA/MRA/DSA
  4. CTA/MRA/DSA confirmed multi-vascular regional occlusion (such as bilateral anterior circulation or anterior/posterior circulation, extracranial carotid artery with intracranial tandem lesions), or clinical evidence of bilateral or multi-regional infarction
  5. CTA/MRA/DSA confirms moyamoya disease or moyamoya syndrome
  6. CT/MRI confirmed a significant midline shift effect
  7. CT/MRI confirms the presence of intracranial tumors (except cerebellar meningioma) CT/MRI confirmed intracranial hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of all adverse events (AEs) and severe adverse events (SAEs) | 72 hours after randomization
  AEs including:
  1. Severe hypothermia with body temperature<32 degree centigrade
  2. Severe hypotension with systolic blood pressure<90mmHg that needs additional support
  3. Any forms of intracranial hemorrhage
  4. Coma
  5. Death within 72h
  6. Respiratory depression defined as respiration rate<8 bpm/min
  7. Extrapyramidal symptoms including Parkinsonism, dystonia, dyskinesia.
  AEs are defined as severe adverse events(SAEs) if severity reaches grade 3-5 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) ver. 5.0.

SECONDARY OUTCOMES:
Scores of National institutes of health stroke scale (NIHSS) | 24 hours after randomization
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating worse neurologic deficit.
Infarct volume | 72 hours after randomization
  Infarct volume is assessed by Computed Tomography and automatically calculated by software.
Plasma proteomics and metabolomics | 24 hours±6 hours
  Proteomics and metabolomics will be performed using patients' plasma. The purpose is to determine what proteins or metabolites are mediated by C+P and correlated with favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Doctor, Study Chair — Capital Medical University
Locations (1):
- Linyi People's Hospital, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Because this study is an exploratory trial of dose-escalation, we want to decide whether to share the drug based on some of the problems and situations found during the study and the subject's personal decision. The purpose is to protect the privacy of the subjects and the implementation of the study.

REFERENCES:
- [Background] Tarahovsky YS, Fadeeva IS, Komelina NP, Khrenov MO, Zakharova NM. Antipsychotic inductors of brain hypothermia and torpor-like states: perspectives of application. Psychopharmacology (Berl). 2017 Jan;234(2):173-184. doi: 10.1007/s00213-016-4496-2. Epub 2016 Dec 8. PMID 27933367
- [Background] Guan L, Guo S, Yip J, Elkin KB, Li F, Peng C, Geng X, Ding Y. Artificial Hibernation by Phenothiazines: A Potential Neuroprotective Therapy Against Cerebral Inflammation in Stroke. Curr Neurovasc Res. 2019;16(3):232-240. doi: 10.2174/1567202616666190624122727. PMID 31232236
- [Background] Guo S, Cosky E, Li F, Guan L, Ji Y, Wei W, Peng C, Geng X, Ding Y. An inhibitory and beneficial effect of chlorpromazine and promethazine (C + P) on hyperglycolysis through HIF-1alpha regulation in ischemic stroke. Brain Res. 2021 Jul 15;1763:147463. doi: 10.1016/j.brainres.2021.147463. Epub 2021 Apr 1. PMID 33811844
- [Background] Guo S, Li F, Wills M, Yip J, Wehbe A, Peng C, Geng X, Ding Y. Chlorpromazine and Promethazine (C+P) Reduce Brain Injury after Ischemic Stroke through the PKC-delta/NOX/MnSOD Pathway. Mediators Inflamm. 2022 Jul 15;2022:6886752. doi: 10.1155/2022/6886752. eCollection 2022. PMID 35873710
- [Background] Tong Y, Elkin KB, Peng C, Shen J, Li F, Guan L, Ji Y, Wei W, Geng X, Ding Y. Reduced Apoptotic Injury by Phenothiazine in Ischemic Stroke through the NOX-Akt/PKC Pathway. Brain Sci. 2019 Dec 15;9(12):378. doi: 10.3390/brainsci9120378. PMID 31847503
- [Background] Jiang Q, Wills M, Geng X, Ding Y. Chlorpromazine and promethazine reduces Brain injury through RIP1-RIP3 regulated activation of NLRP3 inflammasome following ischemic stroke. Neurol Res. 2021 Aug;43(8):668-676. doi: 10.1080/01616412.2021.1910904. Epub 2021 Apr 8. PMID 33829970
- [Background] Han Y, Geng XK, Lee H, Li F, Ding Y. Neuroprotective Effects of Early Hypothermia Induced by Phenothiazines and DHC in Ischemic Stroke. Evid Based Complement Alternat Med. 2021 Jan 18;2021:1207092. doi: 10.1155/2021/1207092. eCollection 2021. PMID 33531913
- [Background] Lv S, Zhao W, Rajah GB, Dandu C, Cai L, Cheng Z, Duan H, Dai Q, Geng X, Ding Y. Rapid Intervention of Chlorpromazine and Promethazine for Hibernation-Like Effect in Stroke: Rationale, Design, and Protocol for a Prospective Randomized Controlled Trial. Front Neurol. 2021 Mar 17;12:621476. doi: 10.3389/fneur.2021.621476. eCollection 2021. PMID 33815250
- [Background] Seners P, Yuen N, Mlynash M, Snyder SJ, Heit JJ, Lansberg MG, Christensen S, Albucher JF, Cognard C, Sibon I, Obadia M, Savatovsky J, Baron JC, Olivot JM, Albers GW; Mismatch Prevalence Investigators. Quantification of Penumbral Volume in Association With Time From Stroke Onset in Acute Ischemic Stroke With Large Vessel Occlusion. JAMA Neurol. 2023 May 1;80(5):523-528. doi: 10.1001/jamaneurol.2023.0265. PMID 36939736